CLINICAL TRIAL: NCT03302637
Title: Oral Microbiome and Pancreatic Cancer: a Prospective Case-Control Study
Brief Title: Oral Microbiome and Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-00721
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Using DNA extracted from oral samples from these cohorts, 16S rRNA genes were amplified and sequenced, followed by assignment of each sequence to a microbial taxa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: subjects with histology-confirmed incident pancreatic cancer, with no prior history of cancer (except non-melanoma skin cancer), a valid consent, and pre-diagnostic oral wash samples.
  Interventions: Other: 16S rRNA gene sequencing assay
- Control: selected by incidence density sampling63 among cohort members who had no cancer prior to selection, provided a valid consent and an oral wash. Controls were frequency matched to cases by cohort, age at cohort entry (5 year), sex, race, and calendar year of cohort entry.
  Interventions: Other: 16S rRNA gene sequencing assay

INTERVENTIONS:
Other: 16S rRNA gene sequencing assay — extraction of genomic DNA from oral samples using the Mobio DNA Isolation Kit. 16S rRNA amplicons covering variable regions V3 to V4 will be generated using primers (347F-5'GGAGGCAGCAGTRRGGAAT'-3' and 803R 5'-CTACCRGGGTATCTAATCC-3')66 incorporating adapters and a sample barcode sequence at PI's lab. Amplicons will be sequenced with the Roche 454 FLX Titanium sequencing system at the NYU genome technology center, following the manufacturer's specifications.

SUMMARY:
This is a prospective population based study to examine the relationship of oral and pancreatic microbiome, and their functions, to pancreatic cancer risk.

The identification of specific oral bacteria and their functional relationship to pancreatic cancer will advance scientific knowledge on the etiology of pancreatic cancer. This could provide a new microbially-based research paradigm, possibly leading to new drug targets for this disease. Second, the oral bacteria may serve as a readily accessible, non-invasive biomarker for subsequent pancreatic cancer risk, which help to identify people at high risk of this disease. Finally, the identified oral bacteria may lead to microbial prophylactic preventions, with antibiotic therapy aimed at eradicating the specific species associated with increased cancer risk or, alternatively, combined with probiotics to introduce species that are associated with a decreased cancer risk. Thus, the study outcomes will lead to actionable means for pancreatic cancer prevention.

DETAILED DESCRIPTION:
A history of periodontal disease and the presence of circulating antibodies to selected oral pathogens have been associated with increased risk of pancreatic cancer; however, direct relationships of oral microbes with pancreatic cancer have not been evaluated in prospective studies. Investigators examine the relationship of oral microbiota with subsequent risk of pancreatic cancer in a large nested case-control study.

ELIGIBILITY:
Inclusion Criteria:

* DNA extracted from oral wash samples from NIH-PLCO and ACS-CPS cohorts

Exclusion Criteria:

-

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 361 incident adenocarcinoma of pancreas and 371 matched controls from two prospective cohort studies, the American Cancer Society Cancer Prevention Study II and the National Cancer Institute Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial.
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 1992-12-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of bacterial taxa will be compared in oral and pancreatic samples. | 4 Years
  For the taxa present at both sites, correlation between the abundance of taxa will be examined between the two sites. To adjust for confounders, multivariate linear regression will be used with abundance of oral taxa (exposure) and that of pancreas taxa (outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Ahn, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States